CLINICAL TRIAL: NCT02890745
Title: EMPOX - A Randomised, Double-blinded, Placebo Controlled Study That Evaluates the Effect of Empagliflozin on Oxidative Stress in Patients With Type 2 Diabetes
Brief Title: The Effect Effect of Empagliflozin on Oxidative Stress in Patients With Type 2 Diabetes
Acronym: EMPOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henrik Enghusen Poulsen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Henrik Enghusen Poulsen, Professor, DMSc, chief physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-100
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Empagliflozin; Oxidative stress; Oxidative nucleic acid modifications; 8-oxo-7,8-dihydro-2'-deoxyguanosine; 8-oxo-7,8-dihydroguanosine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empagliflozin (Experimental): One tablet 25 mg empagliflozin every morning for 14 days
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): One tablet placebo every morning for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin
  Arms: Empagliflozin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of empagliflozin on oxidative stress in patients with type 2 diabetes. The association is examined by comparing the difference in oxidative modifications before and after 14 days treatment with 25 mg empagliflozin compared to placebo treatment. The study is randomised, double-blinded, and placebo controlled. Each treatment group consists of 17 males with type 2 diabetes. Oxidative modifications are measured by urinary excretion of 8-oxo-7,8-dihydro-2'-deoxyguanosine and 8-oxo-7,8-dihydroguanosine. A student t-test will be performed to compare the drug treatment with placebo. The results will be published in a peer-review journal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* HbA1c: 6.5-9.0%
* Capable of understanding oral- and written information
* Caucasian

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 60 mL/hour/1.73 m2
* Currently receiving insulin treatment
* Coronary artery bypass grafting, percutaneous coronary intervention, acute coronary syndrome, stroke, lung embolism, deep vein thrombosis, or transitory cerebral ischemia within 6 months
* Genital infection within 14 days
* Plasma alanine aminotransferase ≥3 times upper normal limit
* Treatment with sodium glucose cotransporter (SGLT) -2 inhibitor within 2 months
* Hyperglycaemic symptoms
* Psychiatric disorder
* Intolerance to empagliflozin or other agents relevant to study
* Non-compliant

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of 8-oxo-7,8-dihydro-2'-deoxyguanosine (nmol/24h) | Change from baseline after fourteen days of intervention
Urinary excretion of 8-oxo-7,8-dihydroguanosine (nmol/24h) | Change from baseline after fourteen days of intervention

SECONDARY OUTCOMES:
Plasma levels of malondialdehyde | Change from baseline after fourteen days of intervention
Plasma levels of iron, ferritin, transferrin and transferrin saturation | Measured at baseline and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Larsen EL, Andersen A, Kjaer LK, Eickhoff MK, Frimodt-Moller M, Persson F, Rossing P, Lykkesfeldt J, Knop FK, Vilsboll T, Rungby J, Poulsen HE. Effects of two- and twelve-weeks sodium-glucose cotransporter 2 inhibition on DNA and RNA oxidation: two randomized, placebo-controlled trials. Free Radic Res. 2023 Feb;57(2):140-151. doi: 10.1080/10715762.2023.2213820. Epub 2023 May 19. PMID 37171199
- [Derived] Larsen EL, Cejvanovic V, Kjaer LK, Vilsboll T, Knop FK, Rungby J, Poulsen HE. The effect of empagliflozin on oxidative nucleic acid modifications in patients with type 2 diabetes: protocol for a randomised, double-blinded, placebo-controlled trial. BMJ Open. 2017 May 9;7(5):e014728. doi: 10.1136/bmjopen-2016-014728. PMID 28490557